CLINICAL TRIAL: NCT03970083
Title: Quantitative Tumor Oxygen Measurements in Cervical Cancer
Brief Title: A Pilot Study of Quantitative Tumor Oxygen Measurements in Cervical Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Martin King, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 17-596
Record Dates: First submitted 2019-05-24; First posted 2019-05-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Gynecologic Cancer; Cervical Cancer
Keywords: Gynecologic Cancer; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oxygen Levels in Tumors: -Quantitative oxygen measurements will be obtained in a single field of view using T1 sequences

SUMMARY:
This research is studying the level of oxygen in tumors during the brachytherapy procedure.

DETAILED DESCRIPTION:
Tumors with low levels of oxygen have been found to be more resistant to standard radiation and chemotherapy treatments. For patients with tumors with low oxygen levels, it is not well known if higher radiation doses can overcome treatment resistance to radiation. Currently, there are limited ways of measuring tumor oxygen levels. The investigators believe that measuring tumor oxygen levels during the brachytherapy procedure will allow the investigators to develop better and improved oxygen measurement techniques, and ultimately improve clinical outcomes for patients, such as better local tumor control.

This research study is a Pilot Study, meaning that this is the first time investigators are examining the oxygen sensor being used. This study is designed to test the oxygen sensor's ability to measure the oxygen levels within the participant's cervical tumor with the aid of magnetic resonance imaging (MRI) scans. MRI scans use magnets to make detailed images of the participant's tumor and the surrounding normal tissues during the brachytherapy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a biopsy-proven diagnosis of cervical cancer for which interstitial brachytherapy is planned as standard treatment
* Age 18 years or older
* ECOG performance status of 2 or less (see Appendix A)
* Patients who have received prior radiation or chemotherapy may be enrolled on this study
* Participant is deemed to be an appropriate candidate for MR-guided brachytherapy by the radiation oncologist and the patient elects to be treated with MR-guided brachytherapy
* Participant provides informed consent for prospective collection of relevant medical records for analysis of clinical outcome and treatment-planning techniques
* Ability to understand and the willingness to sign a written informed consent document. Participant is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow- up

Exclusion Criteria:

* Participants who have a contraindication to MRI identified by the MR procedure screening form, such as a pacemaker, aneurysm clip, inner ear implant, neurostimulator, or other non-MR-compatible device or implant
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients will be women with cervical cancer.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a tumor oxygen measurement from at least 1 oxygen sensor catheter | 2 years

SECONDARY OUTCOMES:
Complete Metabolic Response | 2 years
  Absence of abnormal FDG uptake at the site of abnormal FDG uptake noted on the pre-treatment FDG-PET study
Local Tumor Control | 2 years
  Tumor control within the radiation field
Disease-Specific Survival | 2 Years
  From start of treatment to time of disease progression or death
Overall Survival | 2 years
  From start of treatment until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Martin King, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation